CLINICAL TRIAL: NCT03624738
Title: Femorofemoral Bypass in Redo Cardiac Surgery: A Safe and Effective Operative Technique
Brief Title: Femorofemoral Bypass in Redo Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed mahmoud ahmed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cardiac surgery
Record Dates: First submitted 2018-07-28; First posted 2018-08-10 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Heart Valve Diseases
Keywords: Femoro-femoral bypass
MeSH Terms: conditions — Heart Valve Diseases | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Femorofemoral bypass in redo cardiac surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with redo cardiac surgery 1 (Active Comparator): Procedure: the patients will undergo femorofemoral bypass
  Interventions: Procedure: Procedure
- Patients with redo cardiac surgery 2 (Active Comparator): Procedure: the patients will undergo conventional Aortobicaval cannulation
  Interventions: Procedure: Procedure

INTERVENTIONS:
Procedure: Procedure — Patients with redo cardiac surgery 1: femoral artery-femoral vein cardiopulmonary bypass (CPB) in order to achieve cardiac decompression prior to sternotomy.
  Patients with redo cardiac surgery 2: only conventional aortobicaval cannulation will be used

SUMMARY:
Redo cardiac surgery are becoming more common with a patient population at greater risk. Sternal re-entry poses the hazard of probable injury to vital structures. To minimize the risk associated with sternal re-entry, the investigators adopted the method of establishing femoral artery-femoral vein cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
Redo cardiac surgery are more frequent with a patient population at greater risk. Repeat sternal entry poses the risk of possible injury to vital structures. These include laceration of the myocardium, especially the right ventricle, injury of great vessels or crossing coronary bypass grafts as the internal mammary grafts in particular, or dislodgement of emboli from patent vein grafts. To minimize the risk associated with sternal re-entry, the investigators adopted the method of establishing femoral artery-femoral vein cardiopulmonary bypass (CPB) in order to achieve cardiac drain prior to sternotomy. Also, femorofemoral bypass support the hemodynamics in cases of redo emergency cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* 25-65 years old
* Patients scheduled for repeat open heart surgery with sternotomy
* informed consent has been obtained

Exclusion Criteria:

* Planned off-pump cardiac surgery
* Vascular disease
* previous operation on femoral artery
* under 25 years of age

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-17 (Estimated); Primary Completion 2019-03-28 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
invasive monitoring of arterial blood pressure | Baseline during operation
  suitable systolic arterial blood pressure between 50 and 60 mmHg during cardiopulmonary bypass.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed mahmoud ahmed, Doctor, Principal Investigator — Lecturer of cardiothoracic surgery, Faculty of Medicine, Assiut University, Assiut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaneko T, Vassileva CM, Englum B, Kim S, Yammine M, Brennan M, Suri RM, Thourani VH, Jacobs JP, Aranki S. Contemporary Outcomes of Repeat Aortic Valve Replacement: A Benchmark for Transcatheter Valve-in-Valve Procedures. Ann Thorac Surg. 2015 Oct;100(4):1298-304; discussion 1304. doi: 10.1016/j.athoracsur.2015.04.062. Epub 2015 Jul 21. PMID 26209480
- [Background] Agrifoglio M, Gennari M, Kassem S, Polvani G. Saphenous vein cannulation in re-redo cardiac surgery. J Card Surg. 2012 Nov;27(6):676-7. doi: 10.1111/jocs.12004. Epub 2012 Oct 15. PMID 23061405
- [Background] Knight JL, Cohn LH. Left thoracotomy and femoro-femoral bypass for reoperative revascularization of the posterior coronary circulation. J Card Surg. 1987 Sep;2(3):343-9. doi: 10.1111/j.1540-8191.1987.tb00192.x. PMID 2979983